CLINICAL TRIAL: NCT00869778
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Therapeutic Hepatitis B Vaccine (Mimogen-based) in Treating Chronic Hepatitis B Patients
Brief Title: Phase 2 Trial of Therapeutic Hepatitis B Vaccine (Mimogen-based) for Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing Jiachen Biotechnology Ltd. (Industry)
Collaborators: Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71006.01
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; HBeAg positive; Therapeutic HBV Vaccine; HBV-specific Cytotoxic T Lymphocyte
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- εPA-44 900μg (Experimental): Inject εPA-44 900μg at week 0, 4, 8, 12, 20, 28.
  Interventions: Biological: εPA-44
- εPA-44 600μg+Placebo 300μg (Experimental): Inject εPA-44 600μg+Placebo 300μg at week 0, 4, 8, 12, 20, 28.
  Interventions: Biological: εPA-44; Other: Placebo
- Placebo 900μg (Placebo Comparator): Inject Placebo 900μg at week 0, 4, 8, 12, 20, 28.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: εPA-44 — subcutaneously injection of εPA-44 at week 0, 4, 8, 12, 20, 28.
  Other Names: Therapeutic HBV vaccine
  Arms: εPA-44 600μg+Placebo 300μg; εPA-44 900μg
Other: Placebo — subcutaneously injection of Placebo at week 0, 4, 8, 12, 20, 28.
  Arms: Placebo 900μg; εPA-44 600μg+Placebo 300μg

SUMMARY:
The purpose is to evaluate efficacy and safety of therapeutic Hepatitis B Virus（HBV） vaccine (mimogen-based) treatment in chronic hepatitis B patients and to explore the most effective dosage and provide the rational for optimal dosing schedule.

DETAILED DESCRIPTION:
First stage(0-76 weeks):

Eligible subjects are enrolled and assigned to 3 groups randomly in a 1:1:1 ratio：

1. εPA-44 600μg group：Subcutaneous inject εPA-44 600μg at week 0, 4, 8, 12, 20, 28；Polyene Phosphatidylcholine Capsules will be taken orally beginning in week 28.
2. εPA-44 900μg group：Subcutaneous inject εPA-44 900μg at week 0, 4, 8, 12, 20, 28；Polyene Phosphatidylcholine Capsules will be taken orally beginning in week 28.
3. Placebo control group：Subcutaneous inject empty liposome at week 0, 4, 8, 12, 20, 28；Polyene Phosphatidylcholine Capsules will be taken orally beginning in week 28.

The study cycle consists of screening and enrollment period (week -6-0), treatment period (week 0-28) and follow-up period (week 28-76).

Second stage(76-144 weeks):

In this follow-up stage the trial is open designed, and all the subjects completed the first stage study(0-76 weeks):

1. Subjects with no virological response and no serological response in the first stage , and refuse to continue the this follow-up study, will be provided domestic Adefovir Dipivoxil for one year freely;
2. Subjects with virological response but no serological response/with serological response but no virological response/neither virological nor serological response in the first stage, and be willing to continue the this follow-up study, will be treated by εPA-44 900 μg；
3. Subjects with both virological and serological response, will be followed-up to 144 weeks with no Adefovir Dipivoxil or εPA-44 900 μg treatment.

The definition of response is defined as below:

1. Virological response: HBV DNA<2.93×10∧3IU/ml at 76 weeks;
2. Serological response: serological conversion of HBeAg at 76 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years, male or female
2. Conforms to diagnosis standard of chronic hepatitis B according to"2005 Guideline for Prevention and Treatment of Hepatitis B", (with positive HBsAg for more than 6 months), and HBV-DNA more than 100000 copies/ml;HBeAg (+),HBsAb(-); Alanine aminotransferase（ALT） within 2 to 10 times of ULN (upper limit of normal)
3. HLA-A2 positive
4. Compensatory liver disease having following hematological and biochemical indicators:WBC≥3.5E+9/L; ANC≥1.5E+9/L; PLT≥80E+9/L; Hb≥110g/L; TBil≤1.5ULN; ALB ≥ lower limit of normal value; BUN (Urea)≤upper limit of normal value; Cr≤upper limit of normal value; prothrombin time(PT) elongation≤3 sec; Activated partial thromboplastin time（APTT） within normal value; Fasting blood glucose≤7.0mmol/L
5. TSH within normal value
6. AFP ≤20ng/ml
7. Uses effective contraception for subject with child-bearing potential (including females and female partners of males)
8. Understands and signs ICF approved by EC
9. Willing to comply with the study procedures and complete the study

Exclusion Criteria:

1. Antibody of HAV IgM, HCV, HDV IgM or HEV IgM is positive
2. Antibody of CMV IgM, EBV IgM or HIV is positive
3. Antinuclear antibody titer>1:160
4. Hepatocarcinoma, suspected hepatocarcinoma or hepatic cirrhosis
5. Has any of the following illnesses or has a severe disease inappropriate for participation in the study based on the investigator's judgment, such as: Cardiovascular system: instable or significant cardiovascular illness such as angina pectoris, heart attack of myocardial infarction, congestive heart failure, severe hypertension, significant arrhythmia or abnormal ECG etc.; Respiratory system: bronchiectasis, bronchial asthma, chronic obstructive pulmonary disease, respiratory failure, etc.; Endocrine, metabolism diseases: diabetes mellitus, uncontrolled thyroid diseases, etc.; Others: autoimmune disorder, active tuberculosis, malignancies (e.g.tumor), neuropathic or metal illness history,etc.
6. Has used anti-HBV drug (Interferon, Lamivudine, Adefovir Dipivoxil, Entecavir and Telbivudine) and immunomodulator (Thymic peptide,etc ) 6 months prior to the administration of study medication
7. Has participated in any other drug clinical investigations within the past 3 months
8. Has allergy habitus or has suspected allergy to study drug
9. Female who is in pregnancy, in lactation or planning to become pregnant during the course of the study
10. Has a history of alcohol abuse (Alcohol consumption for more than 5 years, with daily consumption over 40g for males and over 20g for females) and known drug dependence
11. Has a history of organ transplant (except external corneal transplantation and hair transplantation)
12. Any other factors inappropriate for enrollment in the study or study completion in the view of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, Ph.D., Principal Investigator — Hepatitis Institute of Peking University People's Hospital
Locations (15):
- China (15):
  - The PLA Beijing Military General Hospital, Beijing, Beijing Municipality
  - The 2nd Affiliated Hosptial of Harbin Medical University, Harbin, Heilongjiang
  - Renmin Hosptial of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - 81th Hospital of PLA, Nanjing, Jiangsu
  - Jilin University First Hospital, Changchun, Jilin
  - TangDu Hospital, XiAn, Shanxi
  - The First Affiliated Hospital of Xi'An JiaoTong University, Xi’an, Shanxi
  - West China Hospital,SiChuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - 302 Militray Hosptial of China, Beijing
  - Hepatitis Institute of Peking University People's Hospital, Beijing
  - Southwest Hospital, Chongqing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei L, Zhao T, Zhang J, Mao Q, Gong G, Sun Y, Chen Y, Wang M, Tan D, Gong Z, Li B, Niu J, Li S, Gong H, Zou L, Zhou W, Jia Z, Tang Y, Fei L, Hu Y, Shang X, Han J, Zhang B, Wu Y. Efficacy and safety of a nanoparticle therapeutic vaccine in patients with chronic hepatitis B: A randomized clinical trial. Hepatology. 2022 Jan;75(1):182-195. doi: 10.1002/hep.32109. Epub 2021 Dec 8. PMID 34396571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 15 sites in the China. The first participant was screened on 26 March 2009. The last participant observation for the Week 76 analysis was on 09 October 2011
Pre-assignment Details: 1218 participants were screened and 360 were randomized; 360 randomized participants received at least one dose of study drug, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- εPA-44 900μg: Subcutaneous injection of εPA-44 900μg at week 0, 4, 8, 12, 20, 28.
- εPA-44 600μg: Participants subcutaneous injected εPA-44 600μg+Placebo 300μg at week 0, 4, 8, 12, 20, 28.
- Placebo 900μg: Participants subcutaneous injected Placebo 900μg at week 0, 4, 8, 12, 20, 28.
Period: Overall Study
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Started | 120 | 120 | 120
Completed | 108 | 113 | 110
Not Completed | 12 | 7 | 10
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 5
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Protocol Violation | 5 | 3 | 5
Not completed — Unblinding | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- εPA-44 900μg: Inject εPA-44 900μg at week 0, 4, 8, 12, 20, 28.
  εPA-44: Inject εPA-44 900μg/600μg at week 0, 4, 8, 12, 20, 28.
- εPA-44 600μg+Placebo 300μg: Inject εPA-44 600μg+Placebo 300μg at week 0, 4, 8, 12, 20, 28.
  εPA-44: Inject εPA-44 900μg/600μg at week 0, 4, 8, 12, 20, 28.
  Placebo: Inject Placebo 900μg at week 0, 4, 8, 12, 20, 28.
- Placebo 900μg: Inject Placebo 900μg at week 0, 4, 8, 12, 20, 28.
  Placebo: Inject Placebo 900μg at week 0, 4, 8, 12, 20, 28.
- Total: Total of all reporting groups
Arm/Group | εPA-44 900μg | εPA-44 600μg+Placebo 300μg | Placebo 900μg | Total
Number analyzed (Participants) | 120 | 120 | 120 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (7.28) | 26.9 (8.56) | 27.4 (7.30) | 26.8 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 26 | 33 | 95
  Male | 84 | 94 | 87 | 265
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.92 (2.992) | 21.55 (3.004) | 21.99 (2.643) | 21.74 (2.998)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBeAg Seroconversion at Endpoint .
Description: Primary endpoint data were summarised under "End of Study",using the last available post-baseline observation(Last Observation Carried Forward,LOCF)
Time Frame: Endpoint(LOCF), up to 76 Weeks
Population: Intention-To-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | εPA-44 900μg | εPA-44 600μg+Placebo 300μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
percentage of participants | 38.8 | 28.6 | 20.2

2. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at Weeks 12, 28, 32, 40, 52, 64, 76
Description: HBeAg seroconversion=HBeAg loss and presence of hepatitis B e antibody (HBeAb). HBeAg is a hepatitis B viral protein and is an indicator of active viral replication
Time Frame: serology response at week 12, 28, 32, 40, 52, 64, 76
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Groups:
- εPA-44 900μg: Participants subcutaneous injected εPA-44 900μg at week 0, 4, 8, 12, 20, 28.
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
percentage of participants
  Week 12 | 8.6 | 7.6 | 1.7
  Week 28 | 13.8 | 12.6 | 7.6
  Week 32 | 16.4 | 13.4 | 9.2
  Week 40 | 22.4 | 20.2 | 10.9
  Week 52 | 25.9 | 22.7 | 10.9
  Week 64 | 31.9 | 24.4 | 14.3
  Week 76 | 37.9 | 28.6 | 18.5

3. Secondary Outcome: The Proportion of Patients With Serum HBV DNA Load Decrease Equal or Greater Than 1 Log Scale;
Time Frame: week 12, 28, 32, 40, 52, 64, 76
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
percentage of participants
  Week 12 | 29.3 | 33.6 | 27.7
  Week 28 | 42.2 | 48.7 | 39.5
  Week 32 | 50.0 | 55.5 | 45.4
  Week 40 | 49.1 | 55.5 | 47.9
  Week 52 | 48.3 | 53.8 | 36.1
  Week 64 | 54.3 | 61.3 | 43.7
  Week 76 | 62.1 | 64.7 | 55.5

4. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Weeks 12,28,32,40,52,64,76
Time Frame: week 12, 28, 32, 40, 52, 64, 76
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
percentage of participants
  Week 4 | 9.5 | 4.2 | 6.7
  Week 8 | 12.9 | 8.4 | 11.8
  Week 12 | 19 | 10.9 | 13.4
  Week 28 | 32.8 | 20.2 | 20.2
  Week 32 | 32.8 | 29.4 | 18.5
  Week 40 | 39.7 | 31.9 | 26.9
  Week 52 | 36.2 | 33.6 | 21.8
  Week 64 | 44 | 38.7 | 26.9
  Week 76 | 48.3 | 37.8 | 34.5

5. Secondary Outcome: The Proportion of Patients With Both Negative HBeAg and HBeAb;
Time Frame: at week 12, 28, 32, 40, 52, 64, 76.
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
percentage of participants
  Week 12 | 0 | 0 | 0
  Week 28 | 0 | 0 | 0
  Week 32 | 0 | 0 | 0
  Week 40 | 0 | 0 | 0
  Week 52 | 0 | 0 | 0
  Week 64 | 0 | 0 | 0
  Week 76 | 0.9 | 0.8 | 0

6. Secondary Outcome: The Proportion of Patients With Positive Anti-HBe
Time Frame: at week 12, 28, 32, 40, 52, 64, 76.
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
percentage of participants
  Week 12 | 15.5 | 14.3 | 10.9
  Week 28 | 25.9 | 26.1 | 18.5
  Week 32 | 29.3 | 27.7 | 20.2
  Week 40 | 31.0 | 31.1 | 22.7
  Week 52 | 31.0 | 34.5 | 18.5
  Week 64 | 36.2 | 38.7 | 23.5
  Week 76 | 44.0 | 37.0 | 29.4

7. Secondary Outcome: Change From Baseline by Visit for HBeAg Titer
Description: Measuring the change in value of each visit viewpoints HBeAg titers decreased compared with baseline values
Time Frame: at week 12, 28, 32, 40, 52, 64, 76.
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
IU/mL
  Week 12 | 11.5 (1250.38) | -460.2 (2650.77) | -278.7 (1561.74)
  Week 28 | -285.4 (1343.17) | -725.2 (2774.22) | -450.3 (1673.79)
  Week 32 | -339.3 (1442.08) | -768.3 (2778.79) | -471.3 (1692.48)
  Week 40 | -407.4 (1523.68) | -737.6 (2944.83) | -496.8 (1721.17)
  Week 52 | -410.0 (1637.26) | -788.0 (3015.94) | -458.9 (1791.04)
  Week 64 | -271.8 (1267.02) | -822.8 (3124.94) | -563.4 (1800.32)
  Week 76 | -327.5 (1286.44) | -947.4 (3231.94) | -629.3 (1846.07)

8. Secondary Outcome: The Proportion of Patients With Serum HBV DNA Load Decrease Equal or Greater Than 2 Log Scale;
Time Frame: week 12, 28, 32, 40, 52, 64, 76
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
percentage of participants
  Week 12 | 12.9 | 19.3 | 13.4
  Week 28 | 29.3 | 31.1 | 24.4
  Week 32 | 28.4 | 33.6 | 24.4
  Week 40 | 35.3 | 40.3 | 26.1
  Week 52 | 37.9 | 42.9 | 23.5
  Week 64 | 41.4 | 47.9 | 31.1
  Week 76 | 50.0 | 48.7 | 40.3

9. Secondary Outcome: The Proportion of Patients With Serum HBV DNA Level < 29300 IU / ml;
Time Frame: week 12, 28, 32, 40, 52, 64, 76
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
percentage of participants
  Week 12 | 7.8 | 10.9 | 5.9
  Week 28 | 17.2 | 17.6 | 11.8
  Week 32 | 21.6 | 20.2 | 10.1
  Week 40 | 23.3 | 24.4 | 12.6
  Week 52 | 29.3 | 26.9 | 11.8
  Week 64 | 30.2 | 31.1 | 19.3
  Week 76 | 42.2 | 32.8 | 27.7

10. Secondary Outcome: Change From Baseline by Visit for Serum HBV DNA
Description: Measuring the change in value of each visit viewpoints HBV DNA titers decreased compared with baseline values
Time Frame: week 12, 28, 32, 40, 52, 64, 76
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | εPA-44 900μg | εPA-44 600μg | Placebo 900μg
Number analyzed (Participants) | 116 | 119 | 119
IU/mL
  Week 12 | -176000000 (927000000) | -336000000 (1195000000) | -129000000 (293200000)
  Week 28 | -213000000 (919000000) | -362000000 (1217000000) | -172000000 (299000000)
  Week 32 | -226000000 (925700000) | -372000000 (1218000000) | -172000000 (308500000)
  Week 40 | -229000000 (917000000) | -387000000 (1236000000) | -181000000 (322700000)
  Week 52 | -219000000 (917500000) | -373000000 (1263000000) | -140000000 (311600000)
  Week 64 | -229000000 (932100000) | -362000000 (1045000000) | -168000000 (340500000)
  Week 76 | -276000000 (870500000) | -408000000 (1303000000) | -207000000 (350200000)

ADVERSE EVENTS:
Time Frame: Adverse Events After Dosing（0-76week）
Groups:
- εPA-44 900μg: Inject εPA-44 900μg at week 0, 4, 8, 12, 20, 28.
  εPA-44: Inject εPA-44 at week 0, 4, 8, 12, 20, 28.
- εPA-44 600μg+Placebo 300μg: Inject εPA-44 600μg+Placebo 300μg at week 0, 4, 8, 12, 20, 28.
  εPA-44: Inject εPA-44 at week 0, 4, 8, 12, 20, 28.
  Placebo: Inject Placebo at week 0, 4, 8, 12, 20, 28.
- Placebo 900μg: Inject Placebo 900μg at week 0, 4, 8, 12, 20, 28.
  Placebo: Inject Placebo at week 0, 4, 8, 12, 20, 28.
Arm/Group | εPA-44 900μg | εPA-44 600μg+Placebo 300μg | Placebo 900μg
Serious Adverse Events (participants affected / at risk) | 3/120 | 2/120 | 1/120
Other Adverse Events (participants affected / at risk) | 56/120 | 66/120 | 52/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | εPA-44 900μg (N=120) | εPA-44 600μg+Placebo 300μg (N=120) | Placebo 900μg (N=120)
Acute gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Exacerbation of chronic hepatitis B (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinal bronchogenic cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal liver function (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Right leg fibula fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute exacerbation of hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | εPA-44 900μg (N=120) | εPA-44 600μg+Placebo 300μg (N=120) | Placebo 900μg (N=120)
Local injection site reactions (Skin and subcutaneous tissue disorders) | 6 | 13 | 6
Injection site pain (Skin and subcutaneous tissue disorders) | 3 | 4 | 6
Injection site pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 13 | 10 | 9
Nasopharyngitis (Infections and infestations) | 15 | 20 | 13
weakness (General disorders) | 9 | 6 | 5
Diarrhea (Gastrointestinal disorders) | 6 | 5 | 4
Loss of appetite (Metabolism and nutrition disorders) | 2 | 4 | 1
Oropharyngeal pain (Reproductive system and breast disorders) | 4 | 3 | 1
Coughing (Reproductive system and breast disorders) | 1 | 2 | 4
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 | 0 | 2
Female genital infections (Infections and infestations) | 2 | 4 | 1
Upper abdominal pain (Gastrointestinal disorders) | 3 | 4 | 1
Right upper quadrant pain (Gastrointestinal disorders) | 5 | 2 | 0
nausea (Gastrointestinal disorders) | 3 | 4 | 4
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1 | 1
Injection site swelling (Skin and subcutaneous tissue disorders) | 1 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators can't publish articles relevant to the study unless the sponsor permits.